CLINICAL TRIAL: NCT06692270
Title: Tislelizumab as Single-Agent Neoadjuvant Immunotherapy in Resectable Esophageal Squamous Cell Carcinoma: A Single-Arm, Phase II Clinical Study（TISNEOS）
Brief Title: Tislelizumab as Single-Agent Neoadjuvant Immunotherapy in Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TISNEOS
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-11

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg Q3W, D1 ; 2 cycles

SUMMARY:
Tislelizumab in resectable esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤75 years old, male or female;
* T2-3N0-+M0 or T1bN+M0 thoracic esophageal squamous cell carcinoma (as defined in AJCC 8th Edition) with a definite gastroscopic biopsy.
* There is at least one measurable lesion (RECIST1.1 standard);
* ECOG PS 0~1;
* Expected survival ≥ 12 months;
* Newly diagnosed patients who have not received surgery, chemoradiotherapy, targeted therapy, immunotherapy and other treatments before;
* Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment. Male subjects and women of reproductive age must be on contraception within 24 weeks of starting the first study drug and the last study drug.
* The laboratory test value of the patient before medication shall meet the following criteria:

  1. Blood routine: WBC≥3.0 × 109/L; ANC≥1.5 × 109/L; PLT≥100 × 109/L; HGB≥ 9.0g /dL
  2. Liver function: AST≤2.5 × ULN, ALT≤2.5 × ULN, TBIL≤1.5 × ULN
  3. Renal function: Cr≤1.5 × ULN or CrCl ≥50 mL/min
  4. Coagulation function: INR≤1.5, APTT≤1.5 ×ULN;
* Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Esophageal adenocarcinoma was confirmed by histological or cytological pathology;
* Previous T cell co-stimulation or immune checkpoint therapy, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other T cell-targeting drugs;
* A previous or current history of cancer other than esophageal cancer, other than non-melanoma skin cancer that has been treated therapeutically, cervical cancer in situ, or other cancer that has been treated therapeutically and has not shown signs of recurrence for at least 5 years;
* Interstitial lung disease, drug-induced pneumonia, radiation pneumonia requiring steroid treatment or active pneumonia with clinical symptoms or severe lung dysfunction;
* Uncontrolled hypertension with standard treatment (blood pressure not stabilized below < 150/90 mmHg);
* Hereditary bleeding tendency or coagulation dysfunction. There were clinically significant bleeding symptoms or definite bleeding tendencies within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood ++ or above at baseline;
* Have clinical symptoms or diseases of heart that are not well controlled, such as: (1) NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 24 weeks, (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
* Severe infections (CTCAE > Class 2), such as severe pneumonia requiring hospitalization, bacteremia, and infection complications, occurred within 4 weeks prior to the first use of the study drug;
* Patients with clinically uncontrollable third space effusion (such as pleural effusion/pericardial effusion, who do not need to drain the effusion or have no significant increase in effusion after 3 days of stopping drainage can be included in the group);
* Imaging (CT or MRI) shows that the tumor has invaded the major blood vessels, or the investigator determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study;
* A history of immunodeficiency, including HIV testing positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
* Patients with active hepatitis B (defined as positive HBV surface antigen [HBsAg] test result during screening and HBV-DNA test value higher than the upper limit of normal value in the laboratory of the research center) or hepatitis C (defined as positive HCV surface antibody [HCsAb] test result during screening and HCV-RNA positive);
* Those who have allergic reaction to the experimental drug used in this application;
* According to the investigator's judgment, the subjects have other factors that may lead to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Objective Response Rate | At the end of Cycle 2 (each cycle is 21 days)
  Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor